CLINICAL TRIAL: NCT03367988
Title: Effect of Intraoperative and Post-operative Opioids on Persistent Opioid Use in the Surgical Patient
Brief Title: Opioid Free Anesthesia vs. Opioid Anesthesia Techniques.
Acronym: OFA vs OA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00032413
Record Dates: First submitted 2017-10-25; First posted 2017-12-11 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Analgesic Drug Dependence; Colectomy
Keywords: Opioid Dependence; Analagesia; Opioid-free Anesthesia
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: Single Blinded: Study participants will not know what form of anesthesia they are being given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-free Anesthesia (Experimental): Patients will receive no intraoperative narcotics as part of their anesthesia regimen
  Interventions: Drug: Opioid-free Anesthesia
- Opioid Anesthesia (Active Comparator): Patients will receive intraoperative narcotics as part of their anesthesia regimen
  Interventions: Drug: Opioid Anesthesia

INTERVENTIONS:
Drug: Opioid Anesthesia — Doses/concentration of medications/agents used for the anesthetic management of the subjects enrolled in this trial may be adjusted when necessary to provide optimal subject care. Anesthesia will be induced with rocuronium, propofol, intravenous opioids, and other medication(s)/agent(s) at a concentration range/dose(s) based on the clinical need of the subject.
  Depth of anesthesia will be measured with BIS-monitoring and a standard approaching 50% suppression will be maintained throughout the main duration of surgery. Reversal agent will be administered at a post-tetanic count of 1 or 2.
  Anesthesia will be maintained with IV opioids, propofol and/or medication(s)/agent(s), including inhalation anesthetic agents, at a concentration range/dose(s) based on the clinical need of the subject.
  Tracheal extubation will be performed at the end of anesthesia after administration of reversal agent. After extubation, the investigator will determine when the subject is OR discharge ready.
  Arms: Opioid Anesthesia
Drug: Opioid-free Anesthesia — Doses/concentration of medications/agents used for the anesthetic management of the subjects enrolled in this trial may be adjusted when necessary to provide optimal subject care. Acetaminophen 1g will be given prior to induction. Anesthesia will be induced with rocuronium 1mg, propofol 3-6 mg/kg, and succinylcholine 1.5 mg/kg Depth of anesthesia will be measured with BIS-monitoring and a standard approaching 50% suppression will be maintained throughout the main duration of surgery. Reversal agent will be administered at a post-tetanic count of 1 or 2.
  Anesthesia will be maintained with Sevoflurane, Magnesium, Lidocaine, Ketamine, Decadron, Ondansetron, and Ketorolac at a concentration range/dose(s) based on the clinical need of the subject.
  Tracheal extubation will be performed at the end of anesthesia after administration of reversal agent. After extubation, the investigator will determine when the subject is OR discharge ready.
  Arms: Opioid-free Anesthesia

SUMMARY:
A comparison of post-operative opioid use in Laparoscopic Colectomy patients receiving Opioid or Opioid-free Anesthesia.

DETAILED DESCRIPTION:
The study population will be composed of 100 patients total, 50 opioid-free anesthesia laparoscopic colectomy patients and 50 opioid anesthesia laparoscopic colectomy patients at Tampa General Hospital. After consent is obtained patients will be electronically randomized using REDCap in a 1:1 ratio and assigned to a opioid anesthesia or opioid free anesthesia group. Patients will also consent to be asked survey questions preoperatively and be followed for 12 months postoperatively at specific intervals to evaluate pain, satisfaction, and opioid prescription use. This will be done through a data mining platform and service known as REDCap. REDCap is partnered with USF to allow for subject management, data collection and the distribution of surveys via mobile phone. All data collected by REDCap is stored on a HIPPA compliant server. Patients will receive automated push notifications to their mobile phones to fill out surveys regarding their pill usage, pain, and satisfaction for a year or until cessation of opioid use is confirmed. Confirmation of opioid cessation will be performed on a case by case basis by the principal investigator, Dr. Camporesi. In addition to the surveys performed, nausea and pain scores will be collected prospectively from observation in the PACU

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to TGH for laparoscopic colectomy under Dr. Sanchez's care
* Adults aged 18 and older

Exclusion Criteria:

* Patients who are pregnant
* Patients that are not registered within Tampa General Hospital Electronic Medical Records System
* Patients without smart phone capabilities
* Patients younger than 18 years
* Patients older than 80 years
* Patients who cannot speak or read English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory | Once a week for up to 12 months
  a standardized 9 question survey broken into pain severity and pain interference sections. The sections rank various items relating to their respective categorizations of pain on a scale from 0 to 10. The arithmetic mean of each section can then be utilized to determine Severity of pain and impact of pain on daily function during the past week.
Post-surgical opioid prescription use, # of pills used per week | Once a week for up to 12 months
  Weekly pill use for pain management upon discharge

SECONDARY OUTCOMES:
PACU: Pain Scores | 1 - 3 hours
  Visual Analogue Scale (VAS) pain scores every 15 minutes on a 10 centimeter scale. Using a ruler, the score is determined by measuring the distance (cm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater pain intensity. no pain (0 cm), mild pain(1-4.4 cm), moderate pain (4.5-7.4 cm), and severe pain (7.5-10 cm). Normative values are not available. The scale has to be shown to the patient otherwise it is an auditory scale not a visual one.
PACU: Nausea Scores | 1 - 3 hours
  Postoperative Nausea and Vomiting (PONV) every 15 minutes scores (0-4) 0, no nausea; 1, mild nausea ≤ 15 minutes; 2, nausea ≥ 10 minutes; 3, nausea ≥ 5 minutes; 4, vomiting
PACU: Opioid Use in Morphine Equivalents | 1 - 3 hours
  Total ammount of rescue narcotics used in PACU converted to milligram morphine equivalents using CDC guidelines for prescribing Opioids
Patient Satisfaction | 12 months
  Patient treatment satisfaction survey results
Length of Stay | 1- 5 days
  Total length of hospital stay in hours

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Camporesi, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Carroll I, Barelka P, Wang CK, Wang BM, Gillespie MJ, McCue R, Younger JW, Trafton J, Humphreys K, Goodman SB, Dirbas F, Whyte RI, Donington JS, Cannon WB, Mackey SC. A pilot cohort study of the determinants of longitudinal opioid use after surgery. Anesth Analg. 2012 Sep;115(3):694-702. doi: 10.1213/ANE.0b013e31825c049f. Epub 2012 Jun 22. PMID 22729963
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Waljee JF, Li L, Brummett CM, Englesbe MJ. Iatrogenic Opioid Dependence in the United States: Are Surgeons the Gatekeepers? Ann Surg. 2017 Apr;265(4):728-730. doi: 10.1097/SLA.0000000000001904. No abstract available. PMID 27429023
- [Background] Kharasch ED, Brunt LM. Perioperative Opioids and Public Health. Anesthesiology. 2016 Apr;124(4):960-5. doi: 10.1097/ALN.0000000000001012. No abstract available. PMID 26808634
- [Background] Mauermann E, Filitz J, Dolder P, Rentsch KM, Bandschapp O, Ruppen W. Does Fentanyl Lead to Opioid-induced Hyperalgesia in Healthy Volunteers?: A Double-blind, Randomized, Crossover Trial. Anesthesiology. 2016 Feb;124(2):453-63. doi: 10.1097/ALN.0000000000000976. PMID 26655493

DOCUMENTS (2):
  • Study Protocol (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03367988/Prot_001.pdf
  • Informed Consent Form (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03367988/ICF_000.pdf